CLINICAL TRIAL: NCT04134871
Title: Walking for Health: The Feasibility of a Walking Intervention to Increase Physical Activity and Reduce Sedentary Behaviour in People With Severe Mental Illness
Brief Title: Walking for Health: an Intervention to Increase Physical Activity and Reduce Sedentary Behaviour in People With SMI
Acronym: WORtH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/0078
Record Dates: First submitted 2019-09-06; First posted 2019-10-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Mental Illness; Schizophrenia; Bipolar Disorder; Major Depression; Psychosis
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomised to the intervention group will be invited to attend a group education session where they will be given a step counter and activity diary, they will be invited to weekly group walks and fortnightly coaching 1-1 sessions aimed at setting and reviewing goals to increase physical activity and reduce sedentary behaviour
  Interventions: Behavioral: Group walk and one to one coaching
- Control group (No Intervention): Participants randomised to the control group will be given an information leaflet about being more active during a one-off 1-1 consultation.

INTERVENTIONS:
Behavioral: Group walk and one to one coaching — Participants will be invited to attend a group education session, weekly group walks and fortnightly coaching sessions
  Arms: Intervention group

SUMMARY:
People who have a severe mental illness can have poorer physical health and higher mortality rates than the general population. Their medications combined with low levels of physical activity and increased sedentary behaviour can general population and may help people with severe mental illness to be more active.

A previous feasibility study has been conducted in the UK in a large city with positive findings. The current study will be conducted in rural settings in Northern Ireland and Republic of Ireland. The intervention will last 13 weeks. People with Severe Mental Illness will be randomly assigned into one of two groups. Both groups will get information on the benefits of physical activity. In addition, one group will be shown how to use a step counter to measure their steps, be invited to a weekly group walk, and meet their coach every 2 weeks contribute to this. Walking is a good way to increase physical activity in the to see how they are getting on and to support them.

The research team are interested in finding out how willing clinicians are to recruit people into the study, how willing people are to take part, do people then stick with the programme, and if not the reasons for people dropping out. Qualitative findings will explore whether participants feel they benefited from and enjoyed the programme. Findings will be used to investigate the feasibility to conduct a larger trial like this in the future.

ELIGIBILITY:
Inclusion Criteria:

* Inactive adults (Male or Female; aged ≥18 years)
* Diagnosis of any SMI (schizophrenia, psychosis, bipolar disorder and major depression).

Exclusion Criteria:

* Significant movement impairment
* Identified as 'Active' using the GPPAQ screening tool
* Unable to understand English or lack comprehension to understand the purpose of the study and given written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Study recruitment rate | Through study completion, approx. 18 months
  The number of participants recruited to the study in relation to the number of individuals screened along with reasons for exclusion.
Retention of study participants | Through study completion, approx. 18 months
  The number of participants that complete the study intervention versus the number of dropouts will be analysed along with reasons for drop out.
Level of acceptability assessed by semi-structured interviews | Data will be collected from participants at completion of the intervention, approx 3 months.
  Semi-structured interviews will involve gaining information on participants' level of overall satisfaction with the intervention

SECONDARY OUTCOMES:
Change in activity levels | Data will be collected at baseline and at completion of intervention, approx 3 months.
  Participants' activity levels will be measured at baseline and end of intervention
Change in body weight (kilograms) | Data will be collected at baseline and at completion of intervention, approx 3 months.
  Participants' body weight will be measured at baseline and end of intervention
Change in waist circumference (cm) | Data will be collected at baseline and at completion of intervention, approx 3 months.
  Participants' waist circumference will be measured at baseline and end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M McDonough, PhD, Principal Investigator — Ulster University
Locations (3):
- Louth Meath Midlands HSE, Dundalk, Louth, Ireland
- United Kingdom (2):
  - Western HSCT, Omagh, Tyrone
  - Northern HSCT, Antrim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonough SM, Howes SC, Dillon M, McAuley J, Brady J, Clarke M, Clarke M, Lait E, McArdle D, O'Neill T, Wilson I, Niven A, Williams J, Tully MA, Murphy MH, McDonough CM. A study protocol for a randomised controlled feasibility trial of an intervention to increase activity and reduce sedentary behaviour in people with severe mental illness: Walking fOR Health (WORtH) Study. Pilot Feasibility Stud. 2021 Nov 15;7(1):205. doi: 10.1186/s40814-021-00938-5. PMID 34782018